CLINICAL TRIAL: NCT00635297
Title: Percutaneous Vertebroplasty.Study of Refracture Rates After Prophylactic Vertebroplasty of Adjacent Vertebrae
Brief Title: Percutaneous Vertebroplasty: Prophylactic Treatment of Adjacent Vertebra
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with patient recruitement
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Øivind Gjertsen Md Nevroradiologisk avdeling Ullevål universitetssykehus HF, Ullevål universitetssykehus HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 889 VP
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2008-01

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: osteoporosis; vertebroplasty; prophylactic; vertebrae; fracture
MeSH Terms: conditions — Osteoporosis; Spinal Fractures; Fractures, Bone | interventions — Polymethyl Methacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 50 osteoporotic patients with a vertebral insufficiency fracture will receive treatment of the vertebrae with standard vertebroplasty
  Interventions: Procedure: Percutaneous vertebroplasty
- 2 (Experimental): 50 osteoporotic patients with a vertebral insufficiency fracture will receive treatment of the vertebrae with standard vertebroplasty. The adjacent vertebrae will be treated with 3-5 ml of PMMA
  Interventions: Procedure: Percutaneous vertebroplasty

INTERVENTIONS:
Procedure: Percutaneous vertebroplasty — PMMA injection 3-10 milliliter in each treated vertebrae
  Other Names: PMMA

SUMMARY:
Percutaneous vertebroplasty is a treatment for painful osteoporotic compression fractures. Multiple reports have shown as high as 20 % refracturerates in vertebrae adjacent to those that have been treated with percutaneous vertebroplasty.

The purpose of the study is to determine if prophylactic vertebroplasty of unfractured vertebrae adjacent to the treated fractured vertebrae can reduce the rates of refracture in adjacent vertebrae.

ELIGIBILITY:
Inclusion Criteria:

* CT and MRI proven non healed painful osteoporotic compression fracture in the thoracic and lumbar spine.

Exclusion Criteria:

* Infection
* High grade spinal stenosis
* Contraindications to MRI
* Dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Refracture rate based on MRI and CT after 3 months and one year | 3 months and one year

SECONDARY OUTCOMES:
Pain relief after the procedure based on VAS | 3 months and one year

CONTACTS AND LOCATIONS:
Overall Officials: Per Hj Nakstad, Phd, Study Director — Nevroradiologisk avdeling Ullevål Universitetssykehus HF
Locations (1):
- Nevroradiologisk avdeling Ullevål universitetssykehus HF, Oslo, Oslo County, Norway